CLINICAL TRIAL: NCT02874092
Title: Ticagrelor in Methotrexate-Resistant Rheumatoid Arthritis
Acronym: TIMERA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-01003
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Methotrexate (MTX); Ticagrelor
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rheumatoid Arthritis (Active Comparator): -Receiving Methotrexate at stable doses of 10 to 25 mg weekly for at least 12 weeks
  Interventions: Drug: Ticagrelor; Drug: MTX therapy
- Osteoarthritis (Active Comparator): -Diagnosis of osteoarthritis made by physician.
  Interventions: Drug: MTX therapy

INTERVENTIONS:
Drug: Ticagrelor
  Arms: Rheumatoid Arthritis
Drug: MTX therapy

SUMMARY:
This is an open label study to assess the improvement in the Disease Activity Score for 28-joint counts (DAS28) with ticagrelor given at 90 mg twice daily in patients with RA who have active disease despite MTX therapy (as defined by the inclusion/exclusion criteria). There will also be a cross sectional analysis of baseline platelet activity in subjects with rheumatoid arthritis and osteoarthritis. Subjects in the OA cohort will not receive any study medication, and will only have one study visit.

Patients will receive 90 mg ticagrelor orally bid. The patients will receive drug for 30-days. Methotrexate dose will remain stable throughout the study duration.

DETAILED DESCRIPTION:
The two main goals of this study are to demonstrate the heightened cardiovascular risk in RA by comparing platelet activity, inflammation and endothelial function in baseline rheumatoid arthritis versus age- and sex-matched patients with osteoarthritis; and 2) to demonstrate the effect of ticagrelor in rheumatoid arthritis by the pre- and post- measures of clinical RA severity, platelet activity, inflammation and endothelial function in rheumatoid arthritis before and after ticagrelor therapy.

ELIGIBILITY:
Inclusion Criteria

RA cohort

* Receiving MTX at stable doses of 10 to 25 mg weekly for at least 12 weeks
* Have a DAS28 of 3.2 or higher (The level of disease activity is considered to be low if the DAS28 is 3.2 or less) (Prevoo et al., 1995)

OA cohort

* Diagnosis of osteoarthritis made by physician.

Exclusion Criteria:

RA cohort

* History of sensitivity to study medications or any of their excipients
* Previous intolerance to MTX
* Current treatment with antiplatelet therapy
* Absolute indication for anti-platelet therapy
* Need for chronic oral anticoagulant therapy
* Severe hepatic impairment (eg, ascites and/or clinical signs of coagulopathy)
* Renal failure (eGFR <30 or requiring dialysis)
* A known bleeding diathesis, hemostatic or coagulation disorder, or prior major bleeding
* Prior stroke
* Active pathological bleeding
* History of intracranial haemorrhage
* Life expectancy <12 months based on investigator's judgement
* Patients considered to be at risk of bradycardic events (e.g., known sick sinus syndrome or second or third degree atrioventricular [AV)] block) unless already treated with a permanent pacemaker
* Anemia (hematocrit < 27%)
* Platelet count < 100,000/ml
* Concomitant use of strong CYP 3A inhibitors or inducers
* History of thrombocytopenia or neutropenia
* Pregnant or nursing women, or females with a positive pregnancy test at screening
* Females of child bearing potential not using acceptable method of birth control prior to or during study
* Concern for inability of the patient to comply with study procedures and/or follow up (eg, alcohol or drug abuse)

OA cohort:

* History of sensitivity to study medications or any of their excipients
* Current treatment with antiplatelet therapy
* Absolute indication for anti-platelet therapy
* Need for chronic oral anticoagulant therapy
* Severe hepatic impairment (eg, ascites and/or clinical signs of coagulopathy)
* Renal failure (eGFR <30 or requiring dialysis)
* A known bleeding diathesis, hemostatic or coagulation disorder, or prior major bleeding
* Prior stroke
* Active pathological bleeding
* History of intracranial haemorrhage
* Life expectancy <12 months based on investigator's judgement
* Anemia (hematocrit < 27%)
* Platelet count < 100,000/ml
* History of thrombocytopenia or neutropenia
* Pregnant or nursing women, or females with a positive pregnancy test at screening
* Females of child bearing potential not using acceptable method of birth control prior to or during study
* Concern for inability of the patient to comply with study procedures and/or follow up (eg, alcohol or drug abuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Berger, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Rheumatoid Arthritis: -Receiving Methotrexate at stable doses of 10 to 25 mg weekly for at least 12 weeks
  Ticagrelor
  MTX therapy
- Osteoarthritis: -Diagnosis of osteoarthritis made by physician.
  MTX therapy
Period: Overall Study
Arm/Group | Rheumatoid Arthritis | Osteoarthritis
Started | 7 | 2
Completed | 7 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis | Osteoarthritis | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline age was only collected for the 7 RA participants
  years
    number analyzed (Participants) | 7 | 0 | 7
    (all) | 48 (16) |  | 48 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 6 | 0 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score for 28-joint Counts (DAS28)
Description: The DAS28 is a composite score derived from 4 of these measures. This '28' version is a simplification of the original DAS score, which requires 44 joints to be counted. Other versions of the DAS28 allow the CRP to be used instead of the ESR, or the omission of either. To calculate the DAS28 your rheumatologist or specialist nurse will:-
  count the number of swollen joints (out of the 28), count the number of tender joints (out of the 28), take blood to measure the erythrocyte sedimentation rate (ESR) or C reactive protein (CRP), ask you (the patient) to make a 'global assessment of health' (indicated by marking a 10 cm line between very good and very bad).
  These results are then fed into a complex mathematical formula to produce the overall disease activity score. A DAS28 of greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission.
  The total scale range is from 2 to 10, with higher scores indicating more disease activity.
Time Frame: 30 Days
Population: The Osteoarthritis arm was removed; no data was collected for this arm due to low enrollment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 7
score on a scale
  Baseline | 5.7 (0.4)
  30 days | 4.3 (0.8)

2. Secondary Outcome: Visual Analog Scale Disease Activity
Description: The VAS is a psychometric response scale that ranges from "no pain" (0) to "worst pain" (100); patients mark a line on a continuum to indicate how they are feeling. Provides global assessment of RA severity.
Time Frame: 30 Days
Population: The Osteoarthritis arm was removed; no data was collected for this arm due to low enrollment
Measure: Mean (Standard Deviation); unit: Units on VAS scale
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 7
Units on VAS scale
  Baseline | 47 (22)
  30 days | 23 (18)

3. Secondary Outcome: Change in Brachial Artery Diameter
Description: Endothelial function is characterized by flow-mediated vasodilation of the brachial artery, which is measured by comparing the brachial artery diameter at rest the diameter after increased forearm blood flow (reactive hyperemia). Brachial artery reactivity testing (BART) is a noninvasive technique for evaluating endothelial function
Time Frame: Baseline, 30 Days
Population: The Osteoarthritis arm was removed; no data was collected for this arm due to low enrollment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 7
mm
  Baseline | 2.5 (0.9)
  30 days | 2.5 (1.1)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Rheumatoid Arthritis | Osteoarthritis
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 0/7 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT02874092/Prot_SAP_000.pdf